CLINICAL TRIAL: NCT02772978
Title: A Randomized, Double-Blind Study of Neural Circuit Responses to COMT Inhibitors in PPG
Brief Title: Dopamine Responsivity in Gamblers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Responsible Gaming (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 10-03082 UCSF
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Pathological Gambling
Keywords: decision making; impulsivity
MeSH Terms: conditions — Gambling; Impulsive Behavior | interventions — Tolcapone; Sugars

STUDY DESIGN:
Intervention Model Description: This study is a single-group study in which subjects received both placebo and tolcapone in a randomized, double-blind, counterbalanced, within-subject design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tolcapone arm (Active Comparator): This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion
  Interventions: Drug: Tolcapone
- placebo arm (Placebo Comparator): This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone — Tolcapone is in the medication class of catechol-O-methyltransferase (COMT) inhibitors
  Other Names: Tasmar
  Arms: tolcapone arm
Drug: Placebo — A placebo is a tablet or capsule that looks like the study medication (in this case, tolcapone) but does not contain any active ingredients
  Other Names: Sugar pill
  Arms: placebo arm

SUMMARY:
This study deals with how people decide between rewards of different value. The investigators want to understand how the brain's dopamine system impacts this kind of decision making. The investigators will use a medication, tolcapone, which can temporarily affect the dopamine system.

DETAILED DESCRIPTION:
Tolcapone increases the effects of dopamine in the brain. Dopamine is a substance that is normally present in the brain. It may increase body movement and may also change a person's ability to process information. Tolcapone stops one's own naturally-released dopamine from being broken down as quickly. The investigators are interested in learning if tolcapone has positive effects on a person's decisions about rewards.

ELIGIBILITY:
Inclusion Criteria: This behavioral and fMRI study will recruit alcohol drinkers who also participate in gambling activities. Subjects will be selected in an unbiased fashion with respect to gender and ethnicity, as minority representation issues do not interact with any of the hypotheses. To be eligible to participate in the study, the following inclusion criteria must also be met:

1. Subject is a healthy volunteer between 18-50 years of age.
2. Subject is right handed (important for interpreting MRI activity).
3. If female, subject is non-lactating, not pregnant and using a reliable contraception method (i.e. abstinence, intrauterine device, hormonal birth control or barrier method).
4. Subject is able to read and speak English.
5. Subject is a high school graduate.
6. Subject is able and willing to provide written informed consent.
7. Subject is able to understand and follow the instructions of the investigator, and understand all ratings scales.
8. Subject is in good health.

Exclusion Criteria:

• In order to assess potential contraindications to tolcapone, blood will be tested for routine chemistries including white cell count, red cell count, platelet count, hemoglobin, hematocrit, MCV, MCH, MCHC, RDW, neutrophils, lymphocytes, monocytes, eosinophils, and basophils. Additionally, a hepatic screen will assay total protein, albumin, globulin, A/G ratio, bilirubin (total, direct, and indirect), alkaline phosphatase, AST (SGOT), and ALT (SGPT). Elevation of plasma bilirubin, AST (SGOT), ALT (SGPT), or alkaline phosphatase consistent with liver disease will be grounds for subject exclusion. (Note that ongoing monitoring of liver enzymes will not be necessary, as only a single, counterbalanced dose of tolcapone will be administered to each subject.) Subjects will additionally be urine-screened for illicit drug use and screened for alcohol intoxication via breathalyzer. The 7 drug classes detected include cocaine, amphetamine, methamphetamine, benzodiazepines, THC, opiates & oxycodone. These drugs have been chosen due to their possible interaction with tolcapone and possible cognitive and cardiovascular effects. No identifiers will be put on the test cup and it will be read immediately and discarded by the researcher. Similarly, the results of the breathalyzer will be read and then the test will be discarded. No personal identifiers will be associated with the test results. Subjects who test positive for any of these substances, with the exception of THC, will be excluded from further participation in the study. Subjects who have used any psychoactive drugs (except marijuana) within 2 weeks of the start of the study or more than 10 times in the last year will be excluded from participation in the study.

Subjects will also be excluded if they regularly use medications that affect dopamine levels, or will have used these medications within two weeks of tolcapone administration (such as tolcapone, entacapone, or any of the following: levodopa/carbidopa, amantadine, bromocriptine, pergolide, pramipexole, ropinirole, selegeline, isocarboxazid, phenelzine, tranylcypromine, clozapine, olanzapine, quetiapine, risperidone, ziprasidone, aripiprazole, fluphenazine, haloperidol, perphenazine, pimozide, thiothixene, trifluoperazine, loxapine, molindone, chlorpromazine, mesoridazine, thioridazine, dextroamphetamine, dexmethylphenidate, dextroamphetamine, or methylphenidate).

A licensed health care provider will also conduct a brief physical exam. This exam will search for signs of medical illness, including jaundice or abdominal distension associated with liver disease, that would exclude subjects from participating in the study. Subjects with clinically significant medical or psychiatric illnesses requiring treatment as determined by screening blood tests, medical history, and/or physical exam will not be eligible to participate in the study.

Female subjects will also be screened for pregnancy, as the effects of COMT inhibitors during pregnancy are not adequately known and these compounds can appear in breast milk. (Pregnancy is also a contraindication to MRI scanning). Since subjects may not know they are pregnant, all female subjects recruited to participate in the study will be required to have a urine pregnancy test prior to each session of the study. These requirements will not apply to any female subjects who are post-menopausal.

Active use of substances other than alcohol, tobacco, or marijuana, use of alcohol on the day of the meeting as assessed by breathalyzer testing, reported marijuana use in the 48 hours preceding a testing visit, and/or a positive pregnancy test, will be grounds for exclusion.

For subjects participating in the fMRI, we will administer an extensive questionnaire listing contraindications to MRI scanning. Because the MRI scanner attracts certain metals, subjects who may have metallic objects in their bodies will be excluded. As an additional measure of protection, we will use a hand-held metal detector to screen subjects before entering the scanner. Subjects who experience claustrophobia will also be excluded from participating in the MRI scan.

Known allergy or intolerance to tolcapone or use of an investigational drug within 30 days of the screening visit will be grounds for exclusion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kayser, MD, PhD, Principal Investigator — University of California at San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kayser AS, Allen DC, Navarro-Cebrian A, Mitchell JM, Fields HL. Dopamine, corticostriatal connectivity, and intertemporal choice. J Neurosci. 2012 Jul 4;32(27):9402-9. doi: 10.1523/JNEUROSCI.1180-12.2012. PMID 22764248
- [Result] Kayser AS, Vega T, Weinstein D, Peters J, Mitchell JM. Right inferior frontal cortex activity correlates with tolcapone responsivity in problem and pathological gamblers. Neuroimage Clin. 2016 Dec 20;13:339-348. doi: 10.1016/j.nicl.2016.12.022. eCollection 2017. PMID 28066708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the community between June 2014 and September 2015.
Groups:
- Functional MRI Arm - Tolcapone, Then Placebo; Functional MRI Arm - Placebo, Then Tolcapone: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion
  Tolcapone: Tolcapone is in the medication class of catechol-O-methyltransferase (COMT) inhibitors
  Placebo: A placebo is a tablet or capsule that looks like the study medication (in this case, tolcapone) but does not contain any active ingredients
Period: Overall Study
Arm/Group | Functional MRI Arm - Tolcapone, Then Placebo | Functional MRI Arm - Placebo, Then Tolcapone
Started (First participant enrolled) | 10 (First participant enrolled) | 9
Completed (Last participant enrolled) | 9 (Last participant enrolled) | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Functional MRI Arm: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion
  Tolcapone: Tolcapone is in the medication class of catechol-O-methyltransferase (COMT) inhibitors
  Placebo: A placebo is a tablet or capsule that looks like the study medication (in this case, tolcapone) but does not contain any active ingredients
Arm/Group | Functional MRI Arm
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Barratt Impulsiveness Scale, Non-planning Subscale [Mean (Standard Deviation); unit: units on a scale] — The Barratt Impulsiveness, Non-planning subscale score range is 11-44. Lower scores indicate lower impulsivity and higher scores indicate higher impulsivity.
  units on a scale | 25.6 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between the Impulsive Choice Ratio and Baseline Impulsivity, as Measured With the Barratt Impulsiveness Scale, Non-planning Subscale
Description: The presented value represents a correlation. Subjects completed a delay discounting task while functional MRI images were obtained. In this task, subjects made hypothetical choices between a smaller amount of money available sooner, and a larger amount of money available later. Performance on the delay discounting task, as assessed by the impulsive choice ratio, was determined for both the tolcapone and placebo sessions, and the difference between them (tolcapone minus placebo) was calculated. This difference value was then correlated with scores on the Barratt Impulsiveness Scale, non-planning subscale.
Time Frame: 120 minutes after drug ingestion
Population: The outcome for this study was the correlation between the BIS score, non-planning subscale, and the difference in ICR (tolcapone minus placebo). As such, one Arm/Group is presented below.
Measure: Number; unit: Correlation coefficient
Groups:
- Functional MRI Arm (Tolcapone and Placebo): This cognitive science study consists of a single arm in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. Tolcapone is a medication in the class of catechol-O-methyltransferase (COMT) inhibitors. A placebo is a tablet or capsule that looks like the study medication (in this case, tolcapone) but does not contain any active ingredients.
Arm/Group | Functional MRI Arm (Tolcapone and Placebo)
Number analyzed (Participants) | 17
Correlation coefficient | -0.5
Statistical Analysis 1: Comparison: Functional MRI Arm (Tolcapone and Placebo); The comparison group represents the difference in ICR and the baseline impulsiveness scale, non-planning subscale; Test type: Superiority; p = 0.04, Fisher transformation — The threshold for statistical significance was set to p < 0.05

2. Other Pre Specified Outcome: Correlation Between the Difference in ICR (Tolcapone Minus Placebo) and the Difference in Blood Oxygen Level Dependent (BOLD) Signal in the Brain (Tolcapone Minus Placebo)
Description: The presented value represents a correlation. The difference in performance on the delay discounting task was calculated as the change in ICR (tolcapone minus placebo). In addition, the difference in BOLD activity throughout the brain was determined (tolcapone minus placebo).
Time Frame: 120 minutes after drug ingestion
Population: The outcome for this study was the correlation between the difference in the ICR and the difference in BOLD activity (tolcapone minus placebo). As such, one Arm / Group is presented below.
Measure: Number; unit: Correlation coefficient
Arm/Group | Functional MRI Arm (Tolcapone and Placebo)
Number analyzed (Participants) | 17
Correlation coefficient | -0.76
Statistical Analysis 1: Comparison: Functional MRI Arm (Tolcapone and Placebo); Test type: Superiority; p < 0.05, Fisher transformation — The threshold is set to p < 0.05, corrected for multiple comparisons

ADVERSE EVENTS:
Groups:
- Tolcapone Arm: This cognitive science study consists of a single "arm" in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion
  Tolcapone: Tolcapone is in the medication class of catechol-O-methyltransferase (COMT) inhibitors
  Placebo: A placebo is a tablet or capsule that looks like the study medication (in this case, tolcapone) but does not contain any active ingredients.
Arm/Group | Tolcapone Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
Funding constrained the # of participants <= 20. Please see the open access journal article (Kayser et al, Neuroimage Clinical, 2016) for full details related to procedures, results, and conclusions for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No